CLINICAL TRIAL: NCT01759264
Title: An Observational Study of Fecal Calprotectin as Clinical Tool in Monitoring Moderate-to-severe Crohn's Disease on Adalimumab Induction Therapy: a KoRean Experience
Brief Title: An Observational Study of Fecal Calprotectin as Clinical Tool in Monitoring Moderate-to-severe Crohn's Disease on Adalimumab Induction Therapy: a KoRean Experience (FAIR)
Acronym: FAIR
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-974
Record Dates: First submitted 2012-12-28; First posted 2013-01-03 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Crohn's Disease
Keywords: Fecal Calprotectin; Crohn's Disease; Adalimumab
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate-to-severe Crohn's disease: Adalimumab induction therapy participants with moderate-to-severe Crohn's Disease

SUMMARY:
The objective of this observational study was to assess changes in fecal calprotectin levels and its suitability as a monitoring tool in participants with moderate-to-severe Crohn's Disease who were treated with adalimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's Disease participants were defined as:

1. Active luminal, moderate-to-severe Crohn's Disease with Crohn's disease activity index (CDAI) greater than 220, who started Adalimumab treatment in a normal clinical practice setting.
2. Fecal Calprotectin greater than or equal to 150 microgram/g.
3. Ileocolonic or colonic disease, with or without involvement of proximal gastrointestinal areas.

Exclusion Criteria:

1. Disease restricted to proximal (small bowel, gastroduodenal) gastrointestinal tract.
2. Participants who had undergone colectomy other than ileocecal resection.
3. Pregnancy or breast feeding.
4. Contraindication to any anti-tumor necrosis factors (TNF) agent.
5. Any drug dependency.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate-to-severe Crohn's Disease
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SoRa Lee, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate-to-severe Crohn's Disease
Started | 101
Completed | 91
Not Completed | 10
Not completed — Serious Adverse Events (SAEs) | 1
Not completed — Adverse Event | 1
Not completed — Other | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Discontinued Humira Due to Business Trip | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS): Participants who received at least one dose of study drug.
Arm/Group | Moderate-to-severe Crohn's Disease
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.72 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 67
Fecal Calprotectin [Mean (Standard Deviation); unit: microgram/gram]
  Per ITT Set (N=92) | 1799.59 (2275.28)
  Per PP Set (N=83) | 1871.02 (2345.65)

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Fecal Calprotectin Less Than 150 Microgram/Gram
Description: Fecal calprotectin was monitored as a non-invasive surrogate marker measured by enzyme-linked immunosorbent assays. A stool sample was collected at baseline (Week 0) and every follow up visit.
Time Frame: At Week 8 and 12
Population: Intention-to-treat (ITT) population (Participants who received at least one adalimumab induction treatment and were measured for at least one primary endpoint after baseline) and Per-Protocol (PP) population (ITT participants who met inclusion/exclusion criteria and completed the study without any major protocol deviation).
Measure: Number; unit: Percentage of participants
Groups:
- Moderate-to-severe Crohn's Disease (ITT Population); Moderate-to-severe Crohn's Disease (PP Population): Adalimumab induction therapy participants with moderate-to-severe Crohn's Disease
Arm/Group | Moderate-to-severe Crohn's Disease (ITT Population) | Moderate-to-severe Crohn's Disease (PP Population)
Number analyzed (Participants) | 93 | 83
Percentage of participants
  At Week 8 | 21.84 | 20.25
  At Week 12 | 18.82 | 17.07

2. Primary Outcome: Percentage of Participants With Fecal Calprotectin Less Than 150 Microgram/Gram
Description: as for outcome 1
Time Frame: At Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate-to-severe Crohn's Disease (ITT Population) | Moderate-to-severe Crohn's Disease (PP Population)
Number analyzed (Participants) | 93 | 83
Percentage of participants | 16.30 | 13.25

3. Secondary Outcome: Mean Percent Change of Fecal Calprotectin From Baseline
Description: as for outcome 1
Time Frame: Week 4, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Moderate-to-severe Crohn's Disease (ITT Population) | Moderate-to-severe Crohn's Disease (PP Population)
Number analyzed (Participants) | 93 | 83
Percentage
  Percent Change at Week 4 (N=92, 83) | -34.60 (59.85) | -39.28 (58.59)
  Percent Change at Week 8 (N=86, 79) | -43.14 (51.59) | -45.08 (50.32)
  Percent Change at Week 12 (N=85, 82) | -10.49 (147.38) | -22.43 (88.76)

4. Secondary Outcome: Percentage of Participants With Remission of Crohn's Disease
Description: Crohn's Disease Activity Index (CDAI) was a composite index consisting of a weighted scoring of eight disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600, a higher score indicates increased disease severity. Clinical remission was defined as CDAI score less than 150.
Time Frame: At Week 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate-to-severe Crohn's Disease (ITT Population) | Moderate-to-severe Crohn's Disease (PP Population)
Number analyzed (Participants) | 93 | 83
Percentage of participants
  CDAI scores less than 150 at Week 4 | 66.30 | 69.51
  CDAI scores less than 150 at Week 8 | 72.94 | 76.92
  CDAI scores less than 150 at Week 12 | 83.53 | 83.95

5. Secondary Outcome: Percentage of Participants With Clinical Response (CR) Due to Adalimumab Treatment
Description: CR70 and CR100 was a decrease from baseline (Week 0) in CDAI score of 70 and 100 or more points, respectively, a lower score indicating improvement in disease activity.
Time Frame: At Week 4, 8, and 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Moderate-to-severe Crohn's Disease (ITT Population) | Moderate-to-severe Crohn's Disease (PP Population)
Number analyzed (Participants) | 93 | 83
Percentage of participants
  CR70 at Week 4 | 86.96 | 87.80
  CR70 at Week 8 | 89.41 | 92.31
  CR70 at Week 12 | 94.12 | 95.06
  CR100 at Week 4 | 75.00 | 76.83
  CR100 at Week 8 | 85.88 | 88.46
  CR100 at Week 12 | 90.59 | 91.36

ADVERSE EVENTS:
Time Frame: Adverse events leading to discontinuation of adalimumab treatment were collected from signing of informed consent until 12 weeks
Arm/Group | Moderate-to-severe Crohn's Disease
Serious Adverse Events (participants affected / at risk) | 6/99
Other Adverse Events (participants affected / at risk) | 2/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-to-severe Crohn's Disease (N=99)
Abdominal pain (Gastrointestinal disorders) | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate-to-severe Crohn's Disease (N=99)
Abdominal pain (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.